CLINICAL TRIAL: NCT02397525
Title: An Open-Label Study to Evaluate Retreatment With LIPO-202
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Neothetics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LIPO-202-CL-22
Record Dates: First submitted 2015-03-19; First posted 2015-03-25 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Central Abdominal Bulging

ARMS (1):
- LIPO-202 (Experimental)
  Interventions: Drug: LIPO-202

INTERVENTIONS:
Drug: LIPO-202

SUMMARY:
Evaluate the safety of three 8-week courses of treatment with LIPO-202 in non-obese patients who have central abdominal bulging. Efficacy measurements will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* Provided consent
* Healthy male or non-pregnant female subjects
* BMI < 30 kg/m2
* Stable diet and exercise routine
* Central abdominal bulging that is at least "Slight Bulge, Not Flat"

Exclusion Criteria:

* Have had any treatment of the fat around your abdomen, including surgical procedures (tummy tuck, liposuction), injections for fat loss or treatments with devices to reduce fat in your abdomen
* Plan on starting a weight loss or exercise program during the study.
* Be a woman who is pregnant, breast feeding, have had a baby within 6 months and/or not using appropriate birth control.
* Known hypersensitivity to study drugs
* Prior or current enrollment in any Neothetics (formerly Lithera) study involving LIPO-102 or LIPO-202

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Safety: vital signs, physical exams, laboratory tests | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Maria Feldman, Study Director — Neothetics, Inc
Locations (8):
- United States (8):
  - AboutSkin Dermatology, Englewood, Colorado
  - Dermatology Research Institute, LLC, Coral Gables, Florida
  - Gwinnett Clinical Research Center, Inc, Snellville, Georgia
  - Lupo Center for Aesthetic and General Dermatology, New Orleans, Louisiana
  - Bass Plastic Surgery PLLC, New York, New York
  - DermResearch Center of New York, Stony Brook, New York
  - Dermatology Clinical Research Center of San Antonio, San Antonio, Texas
  - Charlottesville Medical Research, Charlottesville, Virginia